CLINICAL TRIAL: NCT04291430
Title: Establishment and Practice of Multi-dimensional Evaluation System for Recanalization of Symptomatic Non-acute Carotid Artery Occlusion
Brief Title: Multi-dimensional Evaluation System for Recanalization of Symptomatic Non-acute Carotid Artery Occlusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY 2019-134-03
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-02

CONDITIONS: Carotid Artery Occlusion
Keywords: Carotid Artery Occlusion; Endovascular treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center, prospective, exploratory, observational, registration study on patients with symptomatic non-acute carotid artery occlusion to initially evaluate the safety and efficacy of endovascular treatment.

DETAILED DESCRIPTION:
Although patients with symptomatic carotid occlusion were primarily treated with medication, the risk of 2-year stroke recurrence was as high as 22.7%. Ipsilateral stroke and hemodynamic decline are independent risk factors for stroke recurrence in patients with carotid artery occlusion. In addition, long-term cerebral hypoperfusion and decreased cerebrovascular reactivity in patients with carotid artery occlusion may lead to cognitive impairment.

At present, the recanalization time window of anterior circulation large vessel occlusive stroke has been extended to 24 hours under certain evaluation approaches. In order to distinguish from the emergency treatment within 24 hours, patients with carotid artery occlusion over 24 hours are collectively referred as non-acute occlusion.

With the maturity of endovascular technique and the advances of interventional devices, endovascular treatment has become a hotspot of clinical research in this field. Case reports have emerged and prospective studies suggest that recanalization of chronic carotid occlusion may improve the cognitive functions. However, the clinical benefit of endovascular treatment for symptomatic non-acute carotid artery occlusion remained controversial.

The purpose of this study is to establish and verify the efficacy of a multi-dimensional evaluation system of endovascular treatment and recanalization of symptomatic non-acute carotid occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form
2. Age: 18-80 years old;
3. Occlusion of the common carotid artery or internal carotid artery (mTICI=0) confirmed by DSA
4. The origin of occlusive segment is from the common carotid artery or the initial segment of the internal carotid artery to the petrous segment and above, and does not exceed the bifurcation of the internal carotid artery (C7 segment). The distal occluded vessels, including the middle cerebral artery, have no severe stenosis or occlusion confirmed by angiography
5. Occlusion over 24 hours (confirmed by imaging or according to the patient's condition change)
6. Ischemic stroke, TIA or progressive visual/cognition impairment associated with occlusion
7. Distinguishable hypoperfusion area indicated by CT perfusion (CBF decrease)

Exclusion Criteria:

1. Target vessel occlusion caused by radiotherapy, vasculitis, moyamoya disease.
2. Any history of intracranial hemorrhage (imaging confirmed or medical record confirmation, except for SWI recorded micro-bleeding) within 3 months.
3. Large core infarction history or index stroke caused by large core infarction (infarct volume >70ml, or exceeding the MCA territory >1/3, or middle cerebral structural shifting)
4. Disabling before index event (mRS>3)
5. History of serious allergy to contrast media (excluding rash), allergic to heparin, aspirin, clopidogrel, statins, metals and anesthetics, or intolerant to general anesthesia
6. Target vessel tortuous or complex vasculature which may cause procedural difficulty
7. Combined with untreated severe coronary artery stenosis or occlusion, untreated intracranial aneurysms, intracranial tumors (other than meningiomas) or any intracranial vascular malformations
8. Gastrointestinal or urinary bleeding, AMI, craniocerebral trauma, major surgery within 30 days
9. Active bleeding constitution or coagulation disease, platelet count < 50 × 10^9 / L
10. Uncontrolled hypertension (systolic blood pressure > 185mmhg), GLU<2.8 mmol/L, GLU>18mmol/L
11. Severe cardiac insufficiency, severe liver injury (AST or ALT more than 3 times of normal value), severe renal insufficiency (creatinine > 177 μ mol / L)， and other late-stage disease
12. Known to have dementia or mental illness, and unable to complete neurological and cognitive assessment
13. Expected survival time<1 year
14. Pregnant or lactating female
15. Included in other studies and in conflict with this study
16. Other special circumstances not suitable for endovascular surgery by consideration of neuro-physician, neurosurgeon, or neurointerventional

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population with symptomatic non-acute carotid artery occlusion confirmed by clinical and imaging assessment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-12-25 (Actual); Primary Completion 2022-12-24 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of ischemic stroke related to target vessels within 12 months after procedure | 12-month after procedure
  Including TIA, minor stroke, moderate stroke, severe stroke and fatal stroke
NIHSS within 12 months after procedure | 12-month after procedure
  NIHSS. The NIH Stroke Scale measures several aspects of brain function, including consciousness, vision, sensation, movement, speech, and language.A certain number of points are given for each of these physical and cognitive functions during a focused neurological examination. A maximal score of 42 represents the most severe and devastating stroke. The level of stroke severity as measured by the NIH stroke scale scoring system:
  0 = no stroke 1-4 = minor stroke 5-15 = moderate stroke 15-20 = moderate/severe stroke 21-42 = severe stroke
mRS within 12 months after procedure | 12-month after procedure
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. (Score Description: 0---No symptoms at all. 1---No significant disability despite symptoms; able to carry out all usual duties and activities. 2---Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance. 3---Moderate disability; requiring some help, but able to walk without assistance. 4--- Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance. 5---Severe disability; bedridden, incontinent and requiring constant nursing care and attention. 6---Dead.
EQ-5D scale within 12 months after procedure | 12-month after procedure
  The EQ-5D essentially consists of two pages: the EQ-5D descriptive system and the EQ-5D visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems (labelled 1-3). The respondent is asked to indicate his / her health state by checking the box against the most appropriate statement in each of the five dimensions. The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine'( score as 100) and 'The worst health you can imagine' (score as 0). This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
MMSE within 12 months after procedure | 12-month after procedure
  The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia. It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document an individual's response to treatment. The MMSE's purpose has been not, on its own, to provide a diagnosis for any particular nosological entity.
MoCA within 12 months after procedure | 12-month after procedure
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment.The MoCA test is a one-page 30-point test administered in approximately 10 minutes. The MoCA assesses: Short term memory/ Visuospatial abilities/ Executive functions/ Attention, concentration and working memory/ Language/ Orientation to time and place.

SECONDARY OUTCOMES:
Technical success rate | Up to 24 hours after procedure
  Defined as the target vessel residual stenosis less than 50% and mTICI grade ≥ 2b
Procedural success rate | Up to 24 hours after procedure
  Defines as the residual stenosis of the target vessel is less than 50%, and the TICI grade is ≥ 2b, and free of peri-procedural complications.
Recurrence rate of ischemic stroke related to culprit vessel within 30 and 90 days after procedure | 30 days and 90days after procedure
  Including TIA, minor stroke, moderate stroke, severe stroke and fatal stroke
Recurrence rate of all ischemic stroke within 30 days, 90days, and 12 months after procedure | 30 days, 90 days and 12 months after procedure
  Including TIA, minor stroke, moderate stroke, severe stroke and fatal stroke
NIHSS within 30 and 90 days after procedure | 30 days and 90days after procedure
  NIHSS. The NIH Stroke Scale measures several aspects of brain function, including consciousness, vision, sensation, movement, speech, and language.A certain number of points are given for each of these physical and cognitive functions during a focused neurological examination. A maximal score of 42 represents the most severe and devastating stroke. The level of stroke severity as measured by the NIH stroke scale scoring system:
  0 = no stroke 1-4 = minor stroke 5-15 = moderate stroke 15-20 = moderate/severe stroke 21-42 = severe stroke
mRS within 30 and 90 days after procedure | 30 days and 90days after procedure
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. (Score Description: 0---No symptoms at all. 1---No significant disability despite symptoms; able to carry out all usual duties and activities. 2---Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance. 3---Moderate disability; requiring some help, but able to walk without assistance. 4--- Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance. 5---Severe disability; bedridden, incontinent and requiring constant nursing care and attention. 6---Dead.
EQ-5D scale within 30 and 90 days after procedure | 30 days and 90days after procedure
  The EQ-5D essentially consists of two pages: the EQ-5D descriptive system and the EQ-5D visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems (labelled 1-3). The respondent is asked to indicate his / her health state by checking the box against the most appropriate statement in each of the five dimensions. The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine'( score as 100) and 'The worst health you can imagine' (score as 0). This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
MMSE within 30 and 90 days after procedure | 30 days and 90days after procedure
  The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia. It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document an individual's response to treatment. The MMSE's purpose has been not, on its own, to provide a diagnosis for any particular nosological entity.
MoCA scale within 30 and 90 days after procedure | 30 days and 90days after procedure
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment.The MoCA test is a one-page 30-point test administered in approximately 10 minutes. The MoCA assesses: Short term memory/ Visuospatial abilities/ Executive functions/ Attention, concentration and working memory/ Language/ Orientation to time and place.
Improvement of cerebral blood flow in the target vessel area showed by CTP within 30 days and 12 months after procedure. | 30 days and 12 month after procedure
  Quantitative analysis by e-Stroke software

OTHER OUTCOMES:
Peri-procedural complications | Before discharge of hospitalisation
  Including: peri-procedural embolism, arterial dissection, vascular perforation, in-stent thrombus, bradycardia and hypotension caused by vagal reflex, post-procedural hyperperfusion syndrome, procedure related low perfusion infarction, etc.
Mortality caused by any stroke within 12 months after procedure | 12 months after procedure
  Cumulative incidence of death caused by any stroke
All-cause mortality within 12 months after procedure | 12 months after procedure
  Cumulative incidence of all-cause death
Any type of intracranial hemorrhage 12 months after procedure | 12 months after procedure
  Including cerebral parenchyma hemorrhage, subarachnoid hemorrhage, intraventricular hemorrhage, etc.
Symptomatic intracranial hemorrhage within 12 months after procedure | 12 months after procedure
  Defined as any type of intracranial hemorrhage resulting in an increase of NIHSS score ≥ 4 or death
The incidence of in-stent restenosis /re-occlusion confirmed by DSA within 12 months after procedure | 12 months after procedure
  Restenosis means that the stenosis in the stent segment, including both ends of the stent, increased by 30% or more than 70% of the residual stenosis immediately after stent implantation; the severity of stenosis was measured using the NASCET standard.
Bailout treatment within 12 months after procedure | 12 months after procedure
  Re-endovascular treatment, carotid endarterectomy or intracranial and extracranial bypass, etc

CONTACTS AND LOCATIONS:
Overall Officials: Dapeng Mo, PhD, Principal Investigator — Beijing Tiantan Hospital; Zhongrong Miao, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China